CLINICAL TRIAL: NCT05020951
Title: Pilot Study to Enable Electronic Laboratory Data Transfer Into Medidata Rave
Brief Title: Pilot Study to Enable Electronic Laboratory Data Transfer From Participating Institutions to MediData/RAVE
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Pediatric Brain Tumor Consortium (Network)
Responsible Party: Sponsor
Other Study IDs: PEPN21EHR; PCTC-N15 (Other: Pediatric Brain Tumor Consortium (PBTC))
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Accurate and Complete Data Acquisition for Clinical Trials

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laboratory Data: Electronic transfer of laboratory data from participating institutions' local electronic health records to the Medidata/RAVE
  Interventions: Other: Medidata RAVE

INTERVENTIONS:
Other: Medidata RAVE — Data collection done exclusively through Medidata Rave. Medidata Rave is a clinical data management system being used for data collection for this trial/study. Access to the trial in Rave is controlled through the CTEP-IAM system and role assignments.

SUMMARY:
An initial step toward more accurate and complete data acquisition for clinical trials, the Pediatric Early Phase Clinical Trials Network (PEP-CTN) and Pediatric Brain Tumor Consortium (PBTC) will assess the feasibility of electronic transfer of laboratory data from participating institutions' local electronic health records to the Medidata/RAVE that is housed within each consortium's Uniform Resource Locator (URL). This study will assess efficiency, effectiveness, and scalability of the laboratory data extraction and transfer processes. This study will identify factors in the process that impact consortium operations, central protocol activation and implementation to the point of declaring the site data-ready.

DETAILED DESCRIPTION:
PRIMARY OBJECITVES

I. To test the feasibility of implementing automated laboratory data extraction and data transfer tools at multiple sites within PEP-CTN and PBTC.

SECONDARY OBJECTIVES

I. To identify and evaluate discrepancies between laboratory data received through retrospective automated laboratory data extraction and manual data ascertainment during the original conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

Patient Data Inclusion Criteria: Specific patient clinical research data to be included in this study for retrospective data capture and analysis will originate from the following PEP-CTN and PBTC studies:

* PEP-CTN: ADVL1412, ADVL1312, ADVL1411
* PBTC: PBTC-042, PBTC-047 (Stratum 1), PBTC-050, PBTC-051 (Stratum 1)

Participating Site Inclusion Criteria: Data from above clinical studies at the following institutions will be included in the initial pilot, with potential to expand to other sites at which patients on these studies were treated.

* Site Participation: Children's Healthcare of Atlanta - Scottish Rite and Egleston, Children's Hospital of Philadelphia, Memorial Sloan Kettering Cancer Center, Seattle Children's Hospital, St. Jude Children's Research Hospital, Texas Children's Hospital, and University of California, San Francisco - Mission Bay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Laboratory data from patients previously enrolled on selected PEP-CTN and PBTC trials. Studies include ADVL1412, ADVL1312, ADVL1411, PBTC-042, PBTC-047 (Stratum 1), PBTC-050, and PBTC-051.
Sampling Method: Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Test the frequency(%) of sites that successfully submitted implementing automated laboratory data extraction and data transfer tools at multiple sites within PEP-CTN and PBTC. | 18 months
  Thorough evaluation of the data extraction and transfer process from each participating site to the PBTC and PEP-CTN databases. Establish feasibility of the proposed process at each site as well as the operations cores.

SECONDARY OUTCOMES:
Identify and evaluate discrepancies between laboratory data received through retrospective automated laboratory data extraction and manual data ascertainment during the original conduct of the study. | 18 months
  Laboratory results identified through automated extraction and transfer will be evaluated to determine if all laboratory results submitted as part of the therapeutic study can be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Miller, MD, MSCE, Study Chair — Children's Healthcare of Atlanta/Emory University
Locations (8):
- United States (8):
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided